CLINICAL TRIAL: NCT03924310
Title: Sensor Glove and Non-Invasive Vibrotactile Feedback Insole to Improve Hand Prostheses Functions and Embodiment
Acronym: FeetBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Berli (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor-Investigator, Martin Berli, Representative of technical orthopedic department, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FeetBack
Record Dates: First submitted 2019-04-15; First posted 2019-04-23 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Amputation; Traumatic, Hand
Keywords: myoelectric prostheses; closed-loop control; vibrotactile feedback; feedback display

STUDY DESIGN:
Intervention Model Description: The two interventions are commercially available myoelectric hand prostheses either with or without an additional feedback device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm amputees (Experimental): This single arm conducts all experiments. In three out of four experiments both interventions (with feedback & without feedback) are used, the fourth experiment does not allow the intervention without feedback.
  Interventions: Device: FeetBack System Active; Device: FeetBack System Passive

INTERVENTIONS:
Device: FeetBack System Active — Commercially available hand prosthesis with feedback device turned on
Device: FeetBack System Passive — Commercially available hand prosthesis with feedback device turned off

SUMMARY:
State-of-the-art myoelectric prostheses provide upper limb amputees with a remarkable variety of grip patterns but lack proper feedback from touch sensation. This restriction limits the controllability of multi-articulated robotic hands, resulting in the rejection of the device in many cases.

Amputees have often reminiscing sensations in the stump, i.e. by touching certain regions, it feels as if no longer existing fingers were touched. These regions form a phantom map and show promising results for touch feedback. However, not every amputee has one and the socket of a prosthesis offers limited space for additional devices. Thus, the investigators developed a feedback display which is worn in the shoe instead of the prosthesis itself. The investigators want to assess the viability of vibrotactile feedback stimulus on the foot as a substitution for pressure on the fingers of an artificial hand in a clinical study. The efforts are based on the hypothesis that a hand prosthesis with tactile feedback has better performance in manipulating fragile and heavy objects, compared with a standard commercial hand prosthesis without tactile feedback.

ELIGIBILITY:
Inclusion Criteria:

* Sign the consent form
* Have basic knowledge of and trust in modern technologies
* Understand the experimental procedures and are willing to participate in the study
* Unilateral below- or above-elbow amputee
* Familiar with the usage of a myoelectric prosthesis

Exclusion Criteria:

* Any form of skin disease
* Contraindication in the device, e.g. hypersensitivity or allergy against materials used in the device
* Impaired condition
* Known or suspected abuse of alcohol or drugs
* Unable to follow the instructions given during the experiments
* Participation at another clinical study with drugs or devices within 30 days before the study at hand
* Homeless person
* Enrollment of the Head of Studies, his/her family members, employees or other dependent persons

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Success rate | Through study completion, an average of 1 month
  Success rate to detect the contact force levels to differentiate between different objects and to manipulate fragile objects, using a hand prosthesis with/without tactile feedback.

SECONDARY OUTCOMES:
Time needed to finish tasks | Through study completion, an average of 1 month
  Comparison of average time needed to finish a set of manipulation tasks, using a hand prosthesis with/without tactile feedback.

OTHER OUTCOMES:
Design acceptance | Up to 2 weeks after study completion
  Design acceptance of the study devices by the subjects with a questionnaire (yes/no, scale, open questions) for further development

CONTACTS AND LOCATIONS:
Overall Officials: Martin Berli, Dr. med., Principal Investigator — Universitätsklinik Balgrist
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Morand R, Brusa T, Schnuriger N, Catanzaro S, Berli M, Koch VM. FeetBack-Redirecting touch sensation from a prosthetic hand to the human foot. Front Neurosci. 2022 Oct 26;16:1019880. doi: 10.3389/fnins.2022.1019880. eCollection 2022. PMID 36389246